CLINICAL TRIAL: NCT07212257
Title: Creation of a Pediatric Reference Database for the Kerpape-Rennes-EMG-Based Gait Index
Acronym: KER-EGI-Kids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles de Kerpape (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-A00178-39
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers; Normal Gait; Child Development; Gait; Normal Gait in Children; Pediatric Normative Gait Data
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy children and adolescents (3-15 years) undergoing gait analysis (Experimental)
  Interventions: Procedure: Gait analysis with surface electromyography (EMG)

INTERVENTIONS:
Procedure: Gait analysis with surface electromyography (EMG) — Each participant undergoes a standardized gait analysis session. After skin preparation, 28 surface electrodes are placed bilaterally on seven lower limb muscles. The child completes 10 walking trials (five round trips of 10 meters) at a comfortable, self-selected speed while being recorded by synchronized cameras. Data collected include Electromyography signals and video recordings. This procedure is non-invasive and performed in a single session lasting approximately one hour

SUMMARY:
Brief Summary

This prospective, monocentric national study aims to establish normative reference data for the Ker-EGI (Kerpape Gait Index), a novel gait quantification index based on muscle activation profiles of the lower limbs in children. The objective is to determine both the mean activation profile and its variability in a healthy pediatric population.

Participants are healthy children and adolescents, aged 3 to 15 years, recruited outside of the Kerpape Rehabilitation Center and specifically attending the Kerpape gait laboratory for this study. A total of 120 subjects are expected. Each participant and their parent(s)/legal guardian provide informed consent prior to enrollment.

Study Procedure:

Each child is accompanied by at least one parent and participates in a single session lasting approximately one hour. After skin preparation (shaving if necessary and cleaning with alcohol), 28 surface electrodes (ECG type) are placed bilaterally on seven lower limb muscles (tibialis anterior, soleus, gastrocnemius medialis, rectus femoris, vastus medialis, semitendinosus, and gluteus medius). Anatomical landmarks are marked with a dermographic pencil. For younger children, a doll is used to facilitate explanation of electrode placement.

The gait analysis is performed with the child in underwear from the time of electrode placement. Each participant completes 10 walking trials (five round trips of 10 meters) at self-selected comfortable speed, following demonstration or a test trial if necessary. Gait is recorded using synchronized cameras and video recordings are anonymized daily.

Data Collection:

Collected data include participant demographics (name, age, sex, height, weight, leg length), electrode signals, and video recordings. Following the session, electrodes are removed, and children are invited to get dressed.

Constraints and Risks:

The study involves a minimal deviation from routine conditions: a single one-hour session including electrode placement, walking assessment, and filming. No invasive procedures or therapeutic interventions are conducted.

Sample Size:

120 healthy children and adolescents, aged 3 to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Child/adolescent aged 3 to 15 years who has given assent, and whose parents (or legal representative) have provided consent to participate in this study.
* Affiliation with a social security system or beneficiary of such a system.

Exclusion Criteria:

* Any known pathology affecting gait pattern (lower limbs, upper limbs, or spine).
* History of orthopedic surgery.
* Behavioral disorder incompatible with data collection.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Normative Kerpape Gait Index-Kids (Ker-EGI Kids) in children | Single session per participant (~1 hour)
  Establishment of a reference database for the Ker-EGI Kids, a gait quantification index based on lower limb muscle activation profiles in children aged 3 to 15 years. The primary outcome is the mean Ker-EGI Kids profile and its variability, with a maximum margin of error of 10%.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles (CMRRF) de Kerpape, Ploemeur, France